CLINICAL TRIAL: NCT01640925
Title: Randomized Controlled Trial of 2% Chlorhexidine Bathing on Nosocomial Infections in the Surgical Intensive Care Unit
Brief Title: Trial of 2% Chlorhexidine Bathing on Nosocomial Infections in the Surgical Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joshua Swan (Other)
Collaborators: Texas Southern University (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Joshua Swan, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00006876; 1211-0239 (Other: HMRI IRB)
Record Dates: First submitted 2012-07-05; First posted 2012-07-16 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Cross Infection; Pneumonia, Ventilator-associated; Catheter-related Infections; Infection Due to Indwelling Urinary Catheter; Surgical Wound Infection
Keywords: nosocomial infection; hospital acquired infection; chlorhexidine; pneumonia, ventilator-associated; catheter-related infections; urinary tract infections, catheter-related; surgical site infection
MeSH Terms: conditions — Cross Infection; Pneumonia, Ventilator-Associated; Catheter-Related Infections; Surgical Wound Infection; Urinary Tract Infections | interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine gluconate bathing (Active Comparator): Upon study enrollment, patients will be bathed with a 2% chlorhexidine gluconate solution on study day 1 and every 48 hours until study completion. The patient will be bathed using standard bathing (non-medicated cloths or soap and water) on study day 2 and every 48 hours after that.
  Interventions: Drug: Chlorhexidine gluconate
- Standard bathing (Placebo Comparator): Upon study enrollment, patients will be bathed using standard bathing (non-medicated cloths or soap and water) daily.
  Interventions: Other: Standard bathing

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Chlorhexidine gluconate 2% solution applied topically for full body bathing once every 48 hours
  Other Names: Bactoshield 4%
  Arms: Chlorhexidine gluconate bathing
Other: Standard bathing — The patient will be bathed using standard bathing (non-medicated cloths or soap and water) daily.
  Arms: Standard bathing

SUMMARY:
This prospective, randomized, controlled trial will compare the incidence of nosocomial infections (composite of primary bloodstream infections, catheter-associated urinary tract infections, ventilator-associated pneumonia, and surgical site infections) that occur in intensive care unit (ICU) patients bathed with 2% chlorhexidine solution versus patients who receive standard bathing (soap and water or non-medicated cloths).

DETAILED DESCRIPTION:
Upon study enrollment, patients will be randomized to one of two study arms. Patients in study arm one will receive standard bathing (soap and water or non-medicated cloth) daily. Patients in study arm two will receive a 2% chlorhexidine bath on study day 1 and every 48 hours and a standard bath (soap and water or non-medicated cloths) on study day 2 and every 48 hours. Patients will be followed until ICU day 28 or discharged from the surgical ICU.

Hypothesis: Compared to standard daily bathing, chlorhexidine-based bathing on ICU admission and every 48 hours will decrease the incidence of nosocomial infections.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the surgical intensive care unit at The Methodist Hospital (Houston, TX)
* Anticipated surgical intensive care unit length of stay of 48 hours or more

Exclusion Criteria:

* Pregnancy
* Age less than 18 years old
* Braden score of less than 9 upon admission to the surgical intensive care unit
* Known allergy to chlorhexidine gluconate
* Active skin irritation upon admission to the surgical intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2012-07; Primary Completion 2013-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua T Swan, Pharm.D., Principal Investigator — The Methodist Hospital, Texas Southern University
Locations (1):
- Surgical Intensive Care Unit, The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data to be determined.

REFERENCES:
- [Result] Swan JT, Bui LN, Pham VP, Shirkey BA, Graviss EA, Hai SA, Ashton CM, Wray NP. "RCT of chlorhexidine versus soap & water bathing for prevention of hospital-acquired infections in SICU". Critical Care Medicine. 2014;42(12 supplement):abstract 4.
- [Result] Swan JT, Ashton CM, Bui LN, Pham VP, Shirkey BA, Blackshear JE, Bersamin JB, Pomer RM, Johnson ML, Magtoto AD, Butler MO, Tran SK, Sanchez LR, Patel JG, Ochoa RA Jr, Hai SA, Denison KI, Graviss EA, Wray NP. Effect of Chlorhexidine Bathing Every Other Day on Prevention of Hospital-Acquired Infections in the Surgical ICU: A Single-Center, Randomized Controlled Trial. Crit Care Med. 2016 Oct;44(10):1822-32. doi: 10.1097/CCM.0000000000001820. PMID 27428384

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chlorhexidine Gluconate Bathing | Standard Bathing
Started | 175 | 175
Completed | 161 | 164
Not Completed | 14 | 11
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Previously enrolled in this trial | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Gluconate Bathing | Standard Bathing | Total
Number analyzed (Participants) | 161 | 164 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (15.9) | 60.2 (16.5) | 59.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 78 | 141
  Male | 98 | 86 | 184

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nosocomial Infection
Description: Proportion of patients with one or more incident nosocomial infections.
  Primary Efficacy Endpoints* (Composite of new nosocomial infection)
  * Primary Bloodstream Infection
  * Catheter Related Urinary Tract Infection
  * Ventilator-Associated Pneumonia**
  * Surgical Site Infection
  (*)Diagnosed using the Centers for Disease Control criteria for hospital acquired infections. Only infections that develop 48 hours or more after study enrollment will be counted as primary endpoints.
  (**)Ventilator associated pneumonia is defined as pneumonia that developed after 48 hours of mechanical ventilation.
Time Frame: Up to 28 days
Measure: Number; unit: participants
Arm/Group | Chlorhexidine Gluconate Bathing | Standard Bathing
Number analyzed (Participants) | 161 | 164
participants | 15 | 30
Statistical Analysis 1: Comparison: Chlorhexidine Gluconate Bathing vs Standard Bathing; Test type: Non-Inferiority or Equivalence — The number of patients needed to achieve 80% power was estimated at 171 using Cox proportional hazards regression (hazard ratio reduction of 0.66; 0.15 probability of infection with control) using a two-sided 5% significance; p = 0.049, Regression, Cox; Cox Proportional Hazard = 0.555, 95% CI 2-sided [0.309 to 0.998] — Hypothesis: Compared to soap and water daily bathing, 2% chlorhexidine gluconate bathing on ICU admission and every 48 hours during surgical ICU care will decrease the risk of acquiring four hospital-acquired infections in surgical ICU patients

2. Secondary Outcome: Incidence of Skin Irritation
Description: The incidence of new onset skin irritation will be recorded and graded for severity using the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03.
Time Frame: up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Bathing | Standard Bathing
Number analyzed (Participants) | 161 | 164
Participants | 30 | 31

3. Secondary Outcome: ICU Length of Stay in Days
Description: Number of days in the ICU after enrollment in study until first ICU discharge.
Time Frame: up to 28 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Chlorhexidine Gluconate Bathing | Standard Bathing
Number analyzed (Participants) | 161 | 164
days | 7.2 (11.4) | 7.0 (8.6)

4. Secondary Outcome: Number of Patients With In-hospital Mortality
Time Frame: up to 28 days or until first hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine Gluconate Bathing | Standard Bathing
Number analyzed (Participants) | 161 | 164
Participants | 22 | 24

ADVERSE EVENTS:
Arm/Group | Chlorhexidine Gluconate Bathing | Standard Bathing
Serious Adverse Events (participants affected / at risk) | 1/161 | 0/164
Other Adverse Events (participants affected / at risk) | 30/161 | 31/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorhexidine Gluconate Bathing (N=161) | Standard Bathing (N=164)
Grade 3 Adverse Skin Occurence (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — One severe (grade 3) skin occurrence was detected in the chlorhexidine arm; however, a blinded reviewer determined that this was due to an allergic reaction to a systemic penicillin antibiotic and was not related to full-body bathing.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chlorhexidine Gluconate Bathing (N=161) | Standard Bathing (N=164)
Incident adverse skin occurrence (Skin and subcutaneous tissue disorders) | 30 (43) | 31 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes